CLINICAL TRIAL: NCT01867645
Title: The Impact of Early Treatment With IgM-enriched IVIG on Critical Illness Polyneuropathy and/or Myopathy in Patients With Multiple Organ Failure and SIRS/Sepsis: A Prospective, Randomized, Placebo-controlled, Double-blinded Trial
Brief Title: The Impact of IVIG Treatment on Critical Illness Polyneuropathy and/or Myopathy in Patients With MOF and SIRS/Sepsis
Acronym: CIPNM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated early due to futility in reaching the primary endpoint.
Sponsor: Medical University of Vienna (Other)
Collaborators: Biotest Pharma GmbH (Unknown); National Bank of Austria (Other Government)
Responsible Party: Principal Investigator, Christian Madl, Univ.-Prof.Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIPNM
Record Dates: First submitted 2013-05-23; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Polyneuropathies
Keywords: Critical illness; Critical illness polyneuropathy and/or myopathy; Intravenous immunoglobulins; Multiple organ failure; SIRS; Sepsis
MeSH Terms: conditions — Polyneuropathies; Critical Illness; Multiple Organ Failure; Sepsis | interventions — Immunoglobulins, Intravenous; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IgM-enriched Intravenous Immunoglobulins (Active Comparator): IgM-enriched IVIG (Pentaglobin, Biotest Pharma GmbH, Dreieich, Germany) at a dose of 0.25g/kg body weight/day as a continuous intravenous infusion at a rate of 2g/h over a period of 3 days
  Interventions: Drug: IgM-enriched Intravenous Immunoglobulins
- Human Albumin (Placebo Comparator): Human albumin 1% (Biotest Pharma GmbH, Dreieich, Germany) as placebo at a dose of 0.25g/kg body weight/day as a continuous intravenous infusion at a rate of 2g/h over a period of 3 days
  Interventions: Drug: Human Albumin

INTERVENTIONS:
Drug: IgM-enriched Intravenous Immunoglobulins — IgM-enriched IVIG (Pentaglobin, Biotest Pharma GmbH, Dreieich, Germany) at a dose of 0.25g/kg body weight/day as a continuous intravenous infusion at a rate of 2g/h over a period of 3 days.
  Other Names: IVIG; IgM-enriched IVIG
  Arms: IgM-enriched Intravenous Immunoglobulins
Drug: Human Albumin — Human albumin 1% (Biotest Pharma GmbH, Dreieich, Germany) as placebo at a dose of 0.25g/kg body weight/day as a continuous intravenous infusion at a rate of 2g/h over a period of 3 days
  Other Names: Placebo
  Arms: Human Albumin

SUMMARY:
Critical illness polyneuropathy and/or myopathy (CIPNM) is a severe complication of critical illness. Retrospective data suggest that early application of IgM-enriched intravenous immunoglobulin (IVIG) may prevent or mitigate CIPNM. Therefore, the primary objective was to assess the effect of early IgM-enriched IVIG versus placebo to mitigate CIPNM in a prospective setting.

DETAILED DESCRIPTION:
Background: Critical illness polyneuropathy and/or myopathy (CIPNM) is a severe complication of critical illness. Retrospective data suggest that early application of IgM-enriched intravenous immunoglobulin (IVIG) may prevent or mitigate CIPNM. Therefore, the primary objective will be to assess the effect of early IgM-enriched IVIG versus placebo to mitigate CIPNM in a prospective setting.

Design: Prospective, randomized, double-blinded and placebo-controlled trial

Setting: Eight-bed medical ICU of a university hospital.

Participants: Critically ill patients will be screened for eligibility defined as multiple organ failure (MOF) and SIRS/sepsis. Patients fulfilling these criteria will be further assessed by a neurologist for clinical signs of CIPNM.

Critically ill patients with multiple organ failure (MOF), SIRS/sepsis, and early clinical signs of CIPNM will be randomized.

ELIGIBILITY:
Inclusion Criteria:

Critically ill patients with failure of at least 2 organ systems diagnosed with SIRS or sepsis fulfilling the following inclusion criteria will be included in this study.

1. Age Range: 18 - 80 years
2. written information and consent as early as possible
3. Male and female patients
4. Clinical signs of incipient CIPNM:

   * decreased tendon reflexes as compared to the admission examination at the ICU
   * or weakness in responsive and co-operative patients as compared to the ad-mission examination at the ICU
   * or signs of incipient muscular atrophy as compared to the admission examination at the ICU

Organ failure:

Patients have to meet at least two of the following 5 criteria:

* cardiovascular system dysfunction: arterial systolic blood pressure<90mm Hg, or mean arterial pressure < 70mm Hg for at least one hour despite adequate fluid resuscitation, adequate intravascular volume status or the use of vasopressors in an attempt to maintain a systolic blood pressure >90mm Hg or a mean arterial pressure >70mm Hg.
* kidney dysfunction: Urine output < 0,5ml/kg body weight/ hour for 1 hour, despite adequate fluid resuscitation
* respiratory system dysfunction: Ratio of PaO2 to FiO2 < 250 in the presence of other dysfunctional organs or systems
* hematologic dysfunction: Platelet count <80.000/mm3 or decreased by 50% in the 3 days preceding enrollment (in the absence of liver cirrhosis or previously known hematological disease)
* metabolic dysfunction: In case of unexplained metabolic acidosis - pH<7,30 or base deficit >5.0mmol/ litre in association with a plasma lactate level >1,5 times of the upper normal limit

SIRS:

Patients have to meet at least three of the following four criteria:

* core temperature >38 or <36°C
* heart rate >90 beats /min, except medical conditions known to increase heart rate
* respiratory rate >20 breaths/min or a PaCO2 of <32mm Hg or the use of mechanical ventilation for an acute respiratory process
* a white- cell count of>12.000 cells/mm3 or <4.000 cells/mm3 or a differential count showing >10% immature neutrophils

Sepsis:

Known or suspected infection evidenced by one or more of the following:

* white cells or bacteria in a normally sterile body fluid
* perforated viscus
* radiographic evidence of pneumonia in the association with the production of purulent sputum
* a syndrome associated with a high risk of infection

Exclusion Criteria:

The inclusion criteria have to be met at the time of enrolment into the study, i.e. at the start of the baseline period. Patients with any of the following conditions will be excluded from the study:

1. Age < 18 years or > 80 years
2. Weight >135 kg
3. Pregnancy or breast-feeding
4. Patients with known absolute IgA-deficiency with proven antibody formation against IgA
5. Patients with known IVIG-intolerability
6. Patients with known pre-existing neuromuscular disorders will not be included. Patients with documented pre-existing severe polyneuropathy will be excluded.
7. Patients with known diseases of the peripheral nerval system and patients with pre-existing disease of the central nerval system with relevant impairment of the motor function.
8. Patients with relevant pulmonary edema secondary to severe heart failure will be excluded because of the relatively high infusion volume (5ml /kg body weight per day over 3 days) determined by the study medication
9. Patients not expected to survive 28 days because of uncorrectable medical condition, such as poorly controlled neoplasma or other end-stage disease
10. Moribund state in which death is perceived to be imminent
11. HIV infection in association with a last known CD4 count of<50/mm3
12. Prediction, based on clinical judgement, that the patient will require chronic ventilatory support for non-respiratory reasons (e.g. neuromuscular disease, paraplegia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-12; Primary Completion 2009-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Effect of early IVIG versus placebo on CIPNM on day 14 | day 14
  The primary outcome was to assess the effect of early IVIG (IgM-enriched Intravenous immunoglobulins) versus placebo to mitigate CIPNM in critically ill patients as assessed by the CIPNM severity sum score on day 14. The CIPNM severity sum score is based on electrophysiological stimulation of the median, ulnar, and tibial nerves on days 0, 4, 7, 14 and on the histological evaluation of muscle biopsies on days 0 and 14 and ranged from 0 (no CIPNM) to 8 (very severe CIPNM).

SECONDARY OUTCOMES:
Effect of early IVIG versus placebo on mortality from any cause within a 28-day period | 28 days
  This secondary outcome aimed to assess the effect of early IVIG versus placebo on mortality from any cause within a 28-day period.
Effect of early IVIG versus placebo on length of the ICU stay. | ICU stay, an expected average of 30 days
  This secondary outcome aimed to assess the effect of early IVIG versus placebo on the length of the ICU stay. Length of ICU stay is defined as the time difference difference between admission of the patient to the ICU and discharge to a (non-ICU) ward or death. This outcome will be assessed an the day of ICU discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Madl, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Brunner R, Rinner W, Haberler C, Kitzberger R, Sycha T, Herkner H, Warszawska J, Madl C, Holzinger U. Early treatment with IgM-enriched intravenous immunoglobulin does not mitigate critical illness polyneuropathy and/or myopathy in patients with multiple organ failure and SIRS/sepsis: a prospective, randomized, placebo-controlled, double-blinded trial. Crit Care. 2013 Oct 2;17(5):R213. doi: 10.1186/cc13028. PMID 24088271